CLINICAL TRIAL: NCT06222905
Title: Analysis of Remote Monitoring / Virtual Clinic Data in Adult Patients With Cystic Fibrosis (CF)
Brief Title: Analysis of Remote Monitoring/Virtual Clinic Data in Adult Patients With Cystic Fibrosis (Project Breathe)
Status: Active, not recruiting | Type: Observational
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Innovate UK (Other Government); Cystic Fibrosis Trust (Other); US Cystic Fibrosis Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: P02445
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: non interventional — non interventional

SUMMARY:
The goal of this observational study is to learn about the impact of home monitoring in adults with cystic fibrosis. The main questions it aims to answer are:

* how people with CF find using home monitoring equipment
* to see if by using home monitoring data acute respiratory exacerbations (chest infections) can be detected earlier than standard care

Participants will be provided with a range of home monitoring equipment -

* hand held spirometer (lung function)
* weighing scales
* oximeter (blood oxygen levels)
* activity and heart rate monitor

to measure health at home several times a week. This information links to an app on a smartphone which the participant and clinicians can see.

DETAILED DESCRIPTION:
This is a multi-centre, observational, prospective cohort study. 610 adult patients with CF will be recruited from the following four CF centres within the United Kingdom

* Royal Papworth Hospital, Cambridge
* University Hospital Llandough, Penarth Wales
* Queen Elizabeth University Hospital, Glasgow, Scotland
* Western General Hospital, Edinburgh, Scotland.

The study is designed to run as a non-disruptive study with no impact on routine clinical practice. Each participant will be actively involved in home monitoring / virtual clinics. linked-anonymised data will be uploaded to a secure National Health Service The approved web-based site for analysis via Microsoft Azure which implements the transmission integrity and confidentiality control by ensuring that cryptography is implemented through a hybrid model.

Clinical metadata including physiology home monitor / virtual clinic data, sputum volume and colour recording will be analysed to establish whether there are predictive signals that could be used as an early alert to clinical deterioration.

Patient level costing will be compared across the cohort and with historical controls to estimate the cost saving or additional cost of home monitoring / virtual clinics.

The statistical data will be analysed by statisticians at the University of Cambridge, with analysis expertise input by Microsoft Research. The health economic data analysis will be carried out by statisticians at the University of Cambridge, with input from the CF Trust and Microsoft Research. A variety of different statistics packages will be utilised as appropriate.

The study specific questionnaire will be completed online by the patients through SurveyMonkey or in paper form if the patient prefers with the questionnaire taking approximately 15 minutes to complete.

All data will be link anonymised and the interviews that take place (at the lead site only) will generate identifiable data, however this will be restricted to the research team at Royal Papworth Hospital and anonymised prior to publication.

Study Duration The study will run for 12 years (with each participant enrolled for up to 5 years (60 months)). The anticipated start date would be 1st December 2018 with the expected end date of the 31 Dec 2030.

Study Activities and Data Collection

The duration of enrolment per participant will be up to 5 years (60 months). During the study period patient data will be collected on the following parameters:

1. Physiology home monitor / virtual clinic data, sputum volume and colour recording metadata will be analysed to establish whether there are predictive signals that could be used as an early alert to clinical deterioration. The above parameters are routinely collected as part of normal clinical care, by using the 'Breathe Remote Monitor which is downloaded onto the patient's own smartphone Patients will need to have access to a Wi-Fi connection, but the app will not create any mobile data charges as long as connected to Wi-Fi.

   The patient can then sync the following devices:

   i. Fitbit - passive monitoring ii. Pulse oximeter - once daily iii. Spirometer - once daily iv. Weighing scales - once daily Anonymised data from the above devices will be uploaded and synced with the app. This will need to be done daily by the patient.
2. Patient level costing data will be compared across the cohort and with historical controls to estimate the cost saving or additional cost of home monitoring / virtual clinics.
3. Semi- structured interviews (at the lead site only) and questionnaires completed through SurveyMonkey or paper (patient can choose) to capture qualitative and quantitative impact of home monitoring / virtual clinics on CF patients. This aspect of the project is the only research procedures that the patients will be asked to undertake.

Patients will be asked to complete the following surveys at the timepoints listed below:

1. Study specific survey completed through either SurveyMonkey or paper copy at 3, 12 and 24 months which will take approximately 15 minutes to complete, no further questionnaires will be required after the first 24 months only the continued collection of data as noted above.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of Cystic Fibrosis based on genetic testing and/or sweat chloride levels
2. Age ≥ 18 years of age
3. Able to provide written informed consent
4. Patients who are known to be suitable for home monitoring and able to manage the process, those currently undertaking home monitoring / virtual clinics

Exclusion Criteria

1. Patients unable to provide written informed consent
2. Patients unwilling to consent to their link anonymized data from home monitoring / virtual clinics being used for research
3. Lung transplant recipients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with cystic fibrosis attending specialist cystic fibrosis centres
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the 12 domain Cystic Fibrosis Questionnaire Revised (CFQR) Score at 24 months | 24 months
  CFQR is a validated, self reported quality of life questionnaire. It has 12 domains such as physical and psychological health. It is a scaled score of 0 to 100. 0 being the worst and 100 the best.

SECONDARY OUTCOMES:
Change from baseline in lung function at 12 months | 12 months
  Lung function (FEV1 % predicted) is a validated measure of lung forced expiratory volume in 1 second.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Floto, Principal Investigator — Royal Papworth Hospital
Locations (2):
- United Kingdom (2):
  - Royal Papworth Hospital, Cambridge, Cambridgeshire
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire

IPD SHARING:
Plan to Share IPD: Undecided